CLINICAL TRIAL: NCT01285232
Title: The Effect of Interleukin-1 Receptor Antagonist on Insulin Secretion in Subjects With Beta Cell Dysfunction
Brief Title: The Effect of Anakinra on Insulin Secretion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: Anakinra1
Record Dates: First submitted 2010-11-08; First posted 2011-01-27 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2010-09

CONDITIONS: Glucose Intolerance; Impaired Insulin Secretion; Diabetes Mellitus Type 2
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2 | interventions — Interleukin 1 Receptor Antagonist Protein; Receptors, Interleukin-6

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anakinra (Experimental): Anakinra 150 mg/day during four weeks
  Interventions: Drug: Anakinra
- Placebo (Placebo Comparator): Placebo during four weeks
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — 150 mg sc once daily during four weeks
  Other Names: Kineret; Interleukin1-receptor antagonist

SUMMARY:
Rationale: Once diabetes develops, β-cell function progressively deteriorates and therapeutic approaches that prevent of delay loss of β-cell function are needed in the treatment of type 2 diabetes mellitus. Recent findings suggest that interleukin-1 (IL-1) may be involved in the progressive β-cell dysfunction in type 2 diabetes mellitus.

Objective: to determine whether blocking IL-1β by recombinant human IL-1ra (anakinra) improves beta-cell function in subjects with β-cell dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Impaired glucose tolerance assessed by oral glucose tolerance test and/or impaired fasting glucose ( ≥ 5.6 mmol/L) and/or HbA1c levels of 5.7-6.4%
* BMI >25 kg/m2
* Age 40-70 years

Exclusion Criteria:

* Known diabetes mellitus
* Fasting plasma glucose ≥ 7.0 mmol/L or HbA1c ≥ 6.5%
* Immunodeficiency or immunosuppressive treatment (including TNFα blocking agents and corticosteroids)
* Use of anti-inflammatory drugs ( including corticosteroids and non steroidal anti-inflammatory drugs, 100 mg or less of aspirin is allowed)
* Signs of current infection (fever, C-reactive protein >30 mmol/L, treatment with antibiotics, previous or current diagnosis of tuberculosis)
* A history of recurrent infections
* Pregnancy or breastfeeding (contraception of at least 3 months before inclusion is required)
* Liver disease defined as aspartate aminotransferase or alanine aminotransferase level of more than three times the upper limit of normal range
* Renal disease defined as MDRD < 60 ml/min/1.73m2
* Neutropenia < 2x 109/L
* Inability to understand the nature and extent of the trial and the procedures required.
* Any medical condition that might interfere with the current study protocol
* Participation in a drug trial within 60 days prior to the first dose

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To determine the effect of anakinra on insulin secretion, as derived from hyperglycemic clamps . | after 4 weeks of treatment with anakinra

SECONDARY OUTCOMES:
To determine the effect on anakinra on insulin sensitivity. | after 4 week treatment of anakinra
  Oral glucose tolerance test
Effects of anakinra on fat cell morphology and gene expression | after 4 weeks of treatment with anakinra
  Fatbiopsy

CONTACTS AND LOCATIONS:
Overall Officials: C.J. Tack, MD, PhD, Prof. of Diabetology, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands